CLINICAL TRIAL: NCT03509545
Title: An Open Label,Crossover Study to Compare Once Daily Dose of 40 mg Torsemide Extended Release to Twice Daily of Furosemide on Natriuresis and Body Weight in Congestive Heart Failure (CHF) Patients Who Are on Stable Dose of Furosemide
Brief Title: Comparison of Once Daily 40 mg Torsemide With Twice-daily 40 mg Furosemide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarfez Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLCD-075-17
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Body Weight Changes
Keywords: natriuresis
MeSH Terms: conditions — Body Weight Changes | interventions — Torsemide; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CHF Patients: ER Torsemide 40 mg (Experimental): CHF patients will be given 40 mg ER Torsemide
  Interventions: Drug: CHF Patients: ER Torsemide 40 mg
- CHF Patients: Furosemide 40 mg (Active Comparator): CHF patients are on 40 mg of Furosemide
  Interventions: Drug: CHF Patients: Furosemide 40 mg

INTERVENTIONS:
Drug: CHF Patients: ER Torsemide 40 mg — ER Torsemide 40mg given once daily to CHF patients
  Other Names: Demadex
  Arms: CHF Patients: ER Torsemide 40 mg
Drug: CHF Patients: Furosemide 40 mg — Stable CHF patients taking twice-daily 40 mg Furosemide
  Other Names: Lasix
  Arms: CHF Patients: Furosemide 40 mg

SUMMARY:
To compare the effects of 40 mg once-daily Torsemide ER to 40 mg twice daily Furosemide on 24-hour sodium excretion.

DETAILED DESCRIPTION:
To compare the effects of 40 mg once-daily Torsemide ER to 40 mg twice-daily Furosemide on changes in body weight after two weeks of treatment. To compare the frequency and volume of urine passed in 24 hours. To compare the patients' quality of life and levels of natriuretic peptide between the two sets of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender over 18 years of age with clinical diagnosis of CHF and on a stable dose of 40 mg Furosemide.

Exclusion Criteria:

* Requirement for any other diuretic, history of cardiac dysrhythmia, other concurrent cardiovascular illness.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
change in 24-hour sodium excretion compared to baseline | 24 hours
  the difference in 24 hour sodium excretion between ER Torsemide and Furosemide

SECONDARY OUTCOMES:
Changes in body weight | 2 weeks
  Body weight changes will be compared between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Anil K, MD, Principal Investigator — Syngene
Locations (1):
- Syngene International, Bangalore, Karnataka, India